CLINICAL TRIAL: NCT03613935
Title: Effect of Changes in Glucose Intake and Sweet Perception on Post Prandial Glycaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 17.19.BIO
Record Dates: First submitted 2018-07-09; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Healthy
MeSH Terms: interventions — LGI4 protein, human

STUDY DESIGN:
Intervention Model Description: This is a monocentric, controlled, randomized, open, complete crossover study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Product 1 (Placebo Comparator): Normal glucose, isosweet, homogeneous: 43 g glucose beverage, with a 43 g glucose equivalent sweetness homogenously delivered
  Interventions: Other: Product 2; Other: Product 3; Other: Product 4
- Product 2 (Active Comparator): Low glucose, isosweet, heterogeneous: 30 g glucose beverage with 43 g glucose equivalent sweetness heterogeneously delivered
  Interventions: Other: Product 1; Other: Product 3; Other: Product 4
- Product 3 (Active Comparator): Low glucose, less sweet, homogeneous: 30 g glucose beverage with a 30 g glucose equivalent sweetness homogenously delivered
  Interventions: Other: Product 1; Other: Product 2; Other: Product 4
- Product 4 (Active Comparator): Low glucose+sucralose, isosweet, homogeneous: 30 g glucose + 18 mg sucralose beverage with a 43 g glucose equivalent sweetness homogenously delivered
  Interventions: Other: Product 1; Other: Product 2; Other: Product 3

INTERVENTIONS:
Other: Product 1 — Comparison with products 2, 3, and 4
  Arms: Product 2; Product 3; Product 4
Other: Product 2 — Comparison with products 1, 3, and 4
  Arms: Product 1; Product 3; Product 4
Other: Product 3 — Comparison with products 1, 2, and 4
  Arms: Product 1; Product 2; Product 4
Other: Product 4 — Comparison with products 1, 2, and 3
  Arms: Product 1; Product 2; Product 3

SUMMARY:
Sugar-sweetened beverages are the main source of added sugars in most Westernized countries, and for this reason constitute a primary target for sugar reduction by many companies, including Nestlé. Instead of using high-intensity sweeteners which are non-caloric in nature, an alternative would be to reduce sugars without altering sweetness.

In this protocol, the general goal is to investigate the relative contribution of sweet taste perception and sugar intake on post-prandial glucose response. 4 different nutritional products will be tested by 16 healthy subjects in a crossover design.

DETAILED DESCRIPTION:
After enrollment, participants will be asked to come to the investigational site 6 times for:

* two sensory tests dedicated to assess the sensory capacity of the participants from the same sensory test repeated twice, for better consistency.
* 4 testing visits for a 3-h blood kinetics after each product intake. These visits will be scheduled on different days separated by a washout period of at least one week. Outcomes will be glycemia and insulinemia.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 29.9 kg/m2
* Fasting capillary blood glucose level ≤ 7 mmol/L
* Able to understand and sign an informed consent form

Exclusion Criteria:

* Pregnancy on anamnesis
* Lactating mothers
* Individuals undergoing either dietary or exercise mediated weight loss program prescribed by a health care professional
* Medically-treated diabetes mellitus or use of anti-hyperglycemic drugs or insulin
* Family history of type 2 diabetes (parents)
* Any other metabolic disease possibly impacting the postprandial glucose and insulin response (to the opinion of the medical doctor)
* Known ageusia or other tasting trouble
* Chronic intake of medications known to affect glucose tolerance to the opinion of the investigator (steroids, protease inhibitors, antidepressants, anxiolytic, or antipsychotics)
* Presence of disease or intake of drug that affects digestion and absorption of nutrients, to the opinion of the medical doctor
* Major medical/surgical event requiring hospitalisation in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Incremental Area under the Curve (iAUC) of plasma glucose | 0 to 3 hours post product intake
  Area under the curve

SECONDARY OUTCOMES:
Incremental Area under the Curve (iAUC) of plasma insulin | 0 to 3 hours post product intake
  Area under the curve
Cmax of plasma glucose | between 0 and 3 hours post product intake
  Maximal concentration of plasma glucose
Cmax of plasma insulin | between 0 and 3 hours post product intake
  Maximal concentration of plasma insulin
Tmax of plasma glucose | between 0 and 3 hours post product intake
  Time (min) for maximal concentration of plasma glucose
Tmax of plasma insulin | between 0 and 3 hours post product intake
  Time (min) for maximal concentration of plasma insulin
Sensory tasting capacity | immediately after product intake
  Assessment of the sweetness of two beverages versus control through a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Beaumont, MD, Principal Investigator — Société des Produits Nestlé (SPN)
Locations (1):
- Nestlé Research Center, Lausanne, Switzerland